CLINICAL TRIAL: NCT05656144
Title: A Single-arm, Single-center, Open-label, Phase II Study Assessing Cadonilimab in the Treatment of Advanced Soft Tissue Sarcoma
Brief Title: Cadonilimab in the Treatment of Advanced Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-006
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab (Experimental): Cadonilimab monotherapy
  Interventions: Device: Cadonilimab

INTERVENTIONS:
Device: Cadonilimab — AK104, 6mg/kg, Q2W

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of Cadonilimab monotherapy in the treatment of patients with advanced soft tissue sarcoma who have received at least one chemotherapy (including anthracyclines) for advanced diseases (excluding alveolar soft part sarcoma).

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a screening period (≤28 days) to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be treated with Cadonilimab monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written and signed informed consent.
* 2. Male or female, age≥ 18 and ≤ 70 years old on day of signing informed consent.
* 3. Pathologically confirmed unresectable or metastatic soft tissue sarcoma, mainly including Undifferentiated pleomorphic sarcoma/malignant fiber histiocytoma, Alveolar soft part sarcoma, dedifferentiated liposarcoma, fibrosarcoma, Leiomyosarcoma, Anigosarcoma, Synovial sarcoma.
* 4. Patients who have failed at least one chemotherapy (including anthracyclines) in the last 6 months (excluding acinar soft tissue sarcoma).

Exclusion Criteria:

* 1. Prior use of investigational products or devices within 4 weeks prior to the first administration of the study treatment.
* 2. Concurrent enrollment into another clinical study, except the study belongs to investigational, non-interventional studies or the follow-up period of interventional studies.
* 3. Prior exposure to any experimental antitumor vaccines, or any agent targeting T-cell costimulation or immune checkpoint pathways (eg, anti-PD-1, anti-PD-L1, anti-CTLA-4, anti-CD137 or anti-OX40 antibody, etc).
* 4. Active autoimmune diseases;
* 5. History of transplantation;
* 6. Known history of primary immunodeficiency virus infection or known history of testing positive for human immunodeficiency virus (HIV).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Anti-tumor activity of Cadonilimab using objective response rate (ORR) based on RECIST v1.1 as assessed by the investigator | up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.

SECONDARY OUTCOMES:
Disease control rate (DCR) | up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1.
Duration of response (DoR) | up to 2 years
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Time to recurrence (TTR) | up to 2 years
  TTR is defined as the time to response base on RECIST v1.1
Progression-free survival (PFS) | up to 2 years
  PFS is defined as the time from the date of first dosing till the first documentation of disease progression (per RECIST v1.1 criteria) or death from any cause (whichever occurs first)
Overall survival (OS) | up to 2 years
  Overall survival is defined as the time from the start of treatment with Cadonilimab until death due to any cause.
AE | From the subject signs the ICF to 30 days (AE) and 90 days (SAE) after the last dose of study treatment or initiation of other anti-tumor therapy, whichever occurs first
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), and clinically significant abnormal laboratory results.